CLINICAL TRIAL: NCT06370728
Title: A Drug-Drug Interaction Study to Assess the Effect of Carbamazepine on the Pharmacokinetics of Orforglipron in Healthy Participants
Brief Title: A Drug-Drug Interaction (DDI) Study of Orforglipron With Carbamazepine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18621; J2A-MC-GZPJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Glucagon-Like Peptide (GLP)- 1
MeSH Terms: interventions — orforglipron; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orforglipron + Carbamazepine (Experimental): Single dose of orforglipron along with twice-daily dose of carbamazepine administered orally
  Interventions: Drug: Orforglipron; Drug: Carbamazepine

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
Drug: Carbamazepine — Administered orally

SUMMARY:
The main purpose of this study is to assess the effect of carbamazepine on the amount of orforglipron in the bloodstream and how long it takes the body to get rid of orforglipron when given orally in healthy study participants. The safety and tolerability of orforglipron and carbamazepine when given separately or together will also be evaluated. The study may last up to approximately 77 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be overtly healthy individuals, assigned male at birth (AMAB) or individuals not of childbearing potential (INOCBP).
* Have a body weight equal to or greater than 45 kg, and body mass index (BMI) between 18.5 and 35.0 kilograms per meter squared (kg/m²), inclusive, at screening.
* Have a hemoglobin level of

  * at least 11.4 g/dL for individuals assigned female at birth (AFAB) and
  * at least 12.5 g/dL for AMAB.
* Have venous access sufficient to allow for blood sampling.

Exclusion Criteria:

* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking orforglipron; or of interfering with the interpretation of data.
* Have an abnormal 12-lead electrocardiogram (ECG).
* Have human leucocyte antigen-B (HLA-B)*1502 or HLA-A*3101 allele; participants with other alleles that demonstrate strong evidence of association with carbamazepine-induced hypersensitivity reaction or hepatic impairment may also be excluded.
* Have a history or presence of multiple or severe allergies, or severe post treatment hypersensitivity reactions.
* Have known allergies to carbamazepine or to orforglipron, related compounds, or any components of the formulation.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC [0-∞]) of Orforglipron | Predose up to Day 18
  PK: AUC (0-∞) of Orforglipron
PK: Area Under the Concentration Versus Time Curve from Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of Orforglipron | Predose up to Day 18
  PK: AUC (0-tlast) of Orforglipron
PK: Maximum Observed Concentration (Cmax) of Orforglipron | Predose up to Day 18
  PK: Cmax of Orforglipron

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No